CLINICAL TRIAL: NCT01434979
Title: Exertional Heat Illness: Biomarkers for Prediction and Return to Duty
Acronym: Heat3
Status: Completed | Type: Observational
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: G191FY
Record Dates: First submitted 2011-09-14; First posted 2011-09-15 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Heat Illness
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Active Duty,DoD Beneficiary, or civilian men and women between the ages of 18 and 45 years, with a waist circumference ≤ 39.4 inches (100 cm) will be asked to participate.
- Exertional Heat Illness / Stroke: Active duty men and women between the ages of 18 and 45 years will be asked to participate. They must have a clinically documented heat stroke within the last year; they will not be tested any sooner than six weeks following the heat stroke. Heat stroke for the purpose of this study is defined as: a syndrome of hyperthermia, physical collapse or debilitation, and encephalopathy as evidenced by delirium, stupor, or coma, occurring during or immediately following exertion or significant heat exposure.

SUMMARY:
The investigators goal is to monitor and quantify the differential physiologic and biomarker responses of controls to standardized exercise under thermoneutral and thermally challenged conditions and responses of exertional heat stroke (EHS) subjects under a thermal-challenged environment to develop unique bio-signature panels to predict those at risk for exertional heat illness (EHI) and guide return to duty following an episode of EHS.

DETAILED DESCRIPTION:
Purpose: Our goal is to monitor and quantify the differential physiologic and biomarker responses of controls to standardized exercise under thermoneutral and thermally challenged conditions and responses of exertional heat stroke (EHS) subjects under a thermal-challenged environment to develop unique biosignature panels to predict those at risk for exertional heat illness (EHI) and guide return to duty following an episode of EHS.

Research Design: This is a prospective cross-sectional study.

Methodology/Technical Approach: The proposed study will examine multiple biomarkers in a group of 100 individuals who have not had an episode of EHS and a prospective study of 50 persons who have had an EHS event. Control subjects will have biomarker assessments before and after an exercise challenge under thermoneutral (TTT) and thermally challenged conditions (heat tolerance test/HTT); differences in the responses to the two tests will be attributed to the heat. In EHS subjects, blood will be obtained at time of injury and then followed up at 6 weeks according to non-EHS controls. In addition, EHS cases will be prospectively followed at 3, 6, 12, and 18 months after the 6-week post assessment. If they are heat tolerant at 6-weeks as determined by a HTT, subsequent measures will include only blood samples and questionnaires, whereas if they are heat intolerant (HIT) at 6-weeks, subsequent measures will include additional HTTs, along with blood samples and questionnaires. As our previous data indicate, approximately 20% of non-EHS persons are HIT; we will test 100 non-EHS and 50 EHI persons in this study. Thus, data will be evaluated with regard to thermotolerance. Importantly, all control participants will undergo two test sessions (HTT and TTT); to control for an order effect, we will randomize the tests.

ELIGIBILITY:
Inclusion Criteria:

* Federal Civilian Employee, Active Duty, or DoD Beneficiary
* Between the ages of 18 and 45 years
* Waist circumference ≤ 39.4 inches (100 cm)
* Willing to walk/run on a treadmill
* Willing to undergo exposure in a thermal chamber
* Willing to maintain their current activity patterns, and to abstain from alcohol, caffeine, and tobacco for 24 hours prior to all sessions
* For cases who have suffered from a exertional heat illness / exertional heat stroke, must have a clinically documented heat stroke within the past year

Exclusion Criteria:

* History of malignant hyperthermia
* Pregnant or lactating
* Have overt heart disease
* Have systolic blood pressure over 140 mm Hg, or diastolic pressure over 90 mm Hg
* Have a waist circumference > 39.4 inches (100 cm)
* Are older than 45 or younger than 18 years of age
* Are anemic
* Are taking psychotropic medication for any mental health disorder
* Are taking other selected medications (glucose lowering, prednisone or beta blockers)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target population will include both civilian DOD beneficiary and active duty military men and women, of any race or ethnicity, between the ages of 18 and 45 years.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2011-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Heat tolerance | 2-hour heat test
  Heat tolerance is determined by physiologic response to a 2-hour heat tolerance test. During this test, participants with core temperature greater than 38.5 C and/or heart rate greater than 150 bpm are considered heat intolerant.

SECONDARY OUTCOMES:
Fitness | 2-hour heat tolerance test
  Body fat and aerobic capacity will be measured to quantify their contribution to heat tolerance.
Behavioral correlates of heat tolerance | past month
  Questionnaires will be used to assess behavioral correlates of heat tolerance, including measures of sleep impairment and executive dysfunction.
Perceived heat strain | 2-hour heat tolerance test and 2-hour control test
  Measures of perceived heat strain will be recorded to determine how accurately participants perceive that they are working in the heat, and whether this adds diagnostic value to the heat test.

OTHER OUTCOMES:
Blood pressure in response to heat tolerance | 2-hour heat tolerance test and 2-hour control test
  Blood pressure will be recorded to see whether it blood pressure response to exercise in the heat correlates with heat tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Deuster, PhD, MPH, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (2):
- Uniformed Services University of the Health Sciences, Bethesda, Maryland, United States
- Heller Institute of Medical Research, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No